CLINICAL TRIAL: NCT03897348
Title: A Pilot Placebo-controlled Human Laboratory Feasibility Study of Lacosamide Effects in Alcohol Use Disorder
Brief Title: Pilot Human Lab Study of Lacosamide in Alcohol Use Disorder (AUD)
Acronym: ACGT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-22180
Record Dates: First submitted 2019-01-02; First posted 2019-04-01 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol craving; human laboratory; lacosamide; non-treatment seeking
MeSH Terms: conditions — Alcoholism | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Crossover Sequence A: Placebo, then Lacosamide 200 mg, then Lacosamide 100 mg (Experimental): Participants receive a single dose of Placebo in ADP Session 1. After a 1 week washout period, they undergo ADP Session 2 in which they receive a single dose of Lacosamide 200 mg. After another 1 week washout period, they undergo ADP Session 3 in which they receive a single dose of Lacosamide 100 mg.
  Interventions: Drug: Placebo; Drug: Lacosamide 100 mg; Drug: Lacosamide 200 mg
- Crossover Sequence B: Lacosamide 200 mg, then Lacosamide 100 mg, then Placebo (Experimental): Participants receive a single dose of Lacosamide 200 mg in ADP Session 1. After a 1 week washout period, they undergo ADP Session 2 in which they receive a single dose of Lacosamide 100 mg. After another 1 week washout period, they undergo ADP Session 3 in which they receive a single dose of Placebo.
  Interventions: Drug: Placebo; Drug: Lacosamide 100 mg; Drug: Lacosamide 200 mg
- Crossover Sequence C: Lacosamide 200 mg, then Placebo, then Lacosamide 100 mg (Experimental): Participants receive a single dose of Lacosamide 200 mg in ADP Session 1. After a 1 week washout period, they undergo ADP Session 2 in which they receive a single dose of Placebo. After another 1 week washout period, they undergo ADP Session 3 in which they receive a single dose of Lacosamide 100 mg.
  Interventions: Drug: Placebo; Drug: Lacosamide 100 mg; Drug: Lacosamide 200 mg
- Crossover Sequence D: Lacosamide 100 mg, then Lacosamide 200 mg, then Placebo (Experimental): Participants receives a single dose of Lacosamide 100 mg in ADP Session 1. After a 1 week washout period, they undergo ADP Session 2 in which they receive a single dose of Lacosamide 200 mg. After another 1 week washout period, they undergo ADP Session 3 in which they receive a single dose of Placebo.
  Interventions: Drug: Placebo; Drug: Lacosamide 100 mg; Drug: Lacosamide 200 mg

INTERVENTIONS:
Drug: Placebo — Oral medication
  Other Names: Placebo capsule identical in appearance to Lacosamide 100 mg and 200 mg capsules.
Drug: Lacosamide 100 mg — Oral medication
  Other Names: Lacosamide 100 mg capsule identical in appearance to Placebo and Lacosamide 200 mg capsule
Drug: Lacosamide 200 mg — Oral medication
  Other Names: Lacosamide 200 mg capsule identical in appearance to Placebo and Lacosamide 100 mg capsules.

SUMMARY:
The overall goal of the proposed project is to improve the treatment of individuals with AUD. The investigators will conduct the first pilot human laboratory study to assess the effects of two doses of lacosamide on alcohol drinking and craving. The investigators will assess its effects on reducing alcohol intake using a human laboratory method, the Yale Alcohol Drinking Paradigm (ADP). The investigators will also assess the feasibility of the Alcohol Drinking Paradigm (ADP) in order to position our research team to have the capacity to conduct future, larger, hypothesis-testing human laboratory-based experiments designed to test the efficacy of potential alcohol treatments.

DETAILED DESCRIPTION:
Four heavy-drinking non-treatment seeking male community volunteers with a diagnosis of AUD will undergo 3 ADP sessions. In each of the 3 ADP sessions, they will receive one of the following 3 different interventions: either 100 mg of lacosamide, 200 mg of lacosamide or placebo.

The ADP session is a one day human laboratory session at the SFVA Medical Center. This human laboratory session involves the self-administration of alcoholic beverages by research participants under highly structured, observed conditions in order to evaluate the effects of the study drug interventions (either 100 mg lacosamide, 200 mg lacosamide, or placebo) on alcohol craving and alcohol consumption. The study follows a double-blind placebo-controlled crossover design in which each participant receives each of the 3 drug interventions in a randomly assigned sequence. There were 4 possible sequences representing the 4 arms of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men, ages 21-50;
2. Able to read English and to complete study evaluations;
3. Meet DSM-V criteria for current alcohol use disorder (AUD);
4. Average weekly alcohol use of 25-70 standard drinks for men over the past 30 days;
5. No more than 3 days/week of alcohol abstinence in the past 30 days, to maximize likelihood that participants will choose to drink during the laboratory sessions.

Exclusion Criteria:

1. Individuals who are seeking AUD treatment or have been in treatment within the past 6 months;
2. Current DSM-V non-alcohol use disorder other than tobacco or cannabis;
3. Positive urine drug test results at more than one baseline appointment for opioids, cocaine, benzodiazepines or barbiturates;
4. Regular use of psychoactive drugs including antipsychotics, anxiolytics and antidepressants during the 30 days prior to entry, as well as anticonvulsants, beta blockers, central nervous system stimulants or depressants, or other drugs that cause excessive sedation;
5. Taking medications that may interact with lacosamide, e.g. medications that prolong the ECG PR interval, or medications with strong CYP3A4 and CYP2C9;
6. Psychosis or any other serious mental illness as judged by SCID and study physician assessment;
7. Medical conditions that in the judgment of the study physician contraindicate the consumption of alcohol;
8. Medical conditions that in the judgment of the study physician contraindicate LAC (non contraindications listed in the FDA-approved Prescribing Information for LAC);
9. Any other medical conditions that in the opinion of the study physician would make study participation hazardous;
10. History of serious alcohol withdrawal (e.g. seizures, DTs, hospitalization) or a Clinical Institute Withdrawal Assessment Scale (CIWA-AD) score greater than or equal to 8;
11. Participants who report disliking spirits will be excluded because 80 proof liquor will be provided during the alcohol self-administration periods;
12. Participants who have taken any investigational drug within 4 weeks preceding study entry;
13. Participants with first-degree atrioventricular block (AV block), PR interval lengthened beyond 0.20 seconds or greater.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — UCSF/SFVAHCS/NCIRE
Locations (1):
- San Francisco VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 participants who were community volunteers were screened for eligibility between September 17, 2018 and April 17, 2019 at the San Francisco VA Medical Center.
Pre-assignment Details: 4 of the 52 were randomized. Of the 48 not randomized, 5 declined to participate and 43 did not meet inclusion criteria.
Period: ADP Session 1
Arm/Group | Crossover Sequence A: Placebo, Then Lacosamide 200 mg, Then Lacosamide 100 mg | Crossover Sequence B: Lacosamide 200 mg, Then Lacosamide 100 mg, Then Placebo | Crossover Sequence C: Lacosamide 200 mg, Then Placebo, Then Lacosamide 100 mg | Crossover Sequence D: Lacosamide 100 mg, Then Lacosamide 200 mg, Then Placebo
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: ADP Session 2
Arm/Group | Crossover Sequence A: Placebo, Then Lacosamide 200 mg, Then Lacosamide 100 mg | Crossover Sequence B: Lacosamide 200 mg, Then Lacosamide 100 mg, Then Placebo | Crossover Sequence C: Lacosamide 200 mg, Then Placebo, Then Lacosamide 100 mg | Crossover Sequence D: Lacosamide 100 mg, Then Lacosamide 200 mg, Then Placebo
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: ADP Session 3
Arm/Group | Crossover Sequence A: Placebo, Then Lacosamide 200 mg, Then Lacosamide 100 mg | Crossover Sequence B: Lacosamide 200 mg, Then Lacosamide 100 mg, Then Placebo | Crossover Sequence C: Lacosamide 200 mg, Then Placebo, Then Lacosamide 100 mg | Crossover Sequence D: Lacosamide 100 mg, Then Lacosamide 200 mg, Then Placebo
Started | 1 | 1 | 0 | 1
Completed | 1 | 1 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Crossover Sequence A: Placebo, Then Lacosamide 200 mg, Then Lacosamide 100 mg: Participant received single dose of placebo in ADP Session 1. After a 1 week washout period, they then underwent ADP Session 2 in which they received a single dose of lacosamide 200 mg. After another 1 week washout period, they underwent ADP Session 3 in which they received a single dose of lacosamide 100 mg.
  (2) 200 mg capsule of lacosamide, an FDA-approved anticonvulsant. A single dose is given at the beginning of 1 of the 3 ADP sessions.
  (3) Placebo. A single dose is given at the beginning of 1 of 3 ADP sessions.
  Lacosamide: Oral medication Placebo: Oral medication
- Crossover Sequence B: Lacosamide 200 mg, Then Lacosamide 100 mg, Then Placebo: Participant received a single dose of lacosamide 200 mg in ADP Session 1. After a 1 week washout period, they then underwent ADP Session 2 in which they received a single dose of lacosamide 100 mg. After another 1 week washout period, they underwent ADP Session 3 in which they received a single dose of placebo.
- Crossover Sequence C: Lacosamide 200 mg, Then Placebo, Then Lacosamide 100 mg: Participant received a single dose of lacosamide 200 mg in ADP Session 1. After a 1 week washout period, they then underwent ADP Session 2 in which they received a single dose of placebo. After another 1 week washout period, they underwent ADP Session 3 in which they received a single dose of lacosamide 100 mg.
- Crossover Sequence D: Lacosamide 100 mg, Then Lacosamide 200 mg, Then Placebo: Participant received a single dose of lacosamide 100 mg in ADP Session 1. After a 1 week washout period, they then underwent ADP Session 2 in which they received a single dose of lacosamide 200 mg. After another 1 week washout period, they underwent ADP Session 3 in which they received a single dose of placebo.
- Total: Total of all reporting groups
Arm/Group | Crossover Sequence A: Placebo, Then Lacosamide 200 mg, Then Lacosamide 100 mg | Crossover Sequence B: Lacosamide 200 mg, Then Lacosamide 100 mg, Then Placebo | Crossover Sequence C: Lacosamide 200 mg, Then Placebo, Then Lacosamide 100 mg | Crossover Sequence D: Lacosamide 100 mg, Then Lacosamide 200 mg, Then Placebo | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 0 | 0 | 1 | 1 | 2
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility (Time, in Months,) Required to Recruit, Screen and Conduct the Study Procedures
Description: Recruitment feasibility will be measured as the time (in months) required to recruit, screen and conduct the study procedures for a total of 4 participants.
Time Frame: 7 months
Measure: Number; unit: months
Arm/Group | Total
Number analyzed (Participants) | 4
months | 7.0

2. Primary Outcome: Retention Feasibility (Proportion of Participants Completing the Alcohol Drinking Paradigm (ADP) Sessions)
Description: Retention feasibility will be measured by the proportion of participants completing the Alcohol Drinking Paradigm (ADP) Sessions 1, 2 and 3.
Time Frame: 6.5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 4
Participants | 3

3. Primary Outcome: Tolerability (Number of Participants With Mild, Moderate, or Severe Adverse Events)
Description: Tolerability will be measured by the number of participants with mild, moderate, and severe adverse events for each of the 3 drug interventions (100 mg lacosamide, 200 mg lacosamide and placebo).
Time Frame: 3 days (1 day each for ADP Session 1, 2, and 3)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: A matching capsule of placebo. A single dose is given at the beginning of 1 of the 3 ADP sessions.
  Placebo: Oral medication
- Lacosamide 100 mg: 100 mg capsule of lacosamide, an FDA-approved anticonvulsant. A single dose is given at the beginning of 1 of the 3 ADP sessions.
  Lacosamide: Oral medication
- Lacosamide 200 mg: 200 mg capsule of lacosamide, an FDA-approved anticonvulsant. A single dose is given at the beginning of 1 of the 3 ADP sessions.
  Lacosamide: Oral medication
Arm/Group | Placebo | Lacosamide 100 mg | Lacosamide 200 mg
Number analyzed (Participants) | 4 | 3 | 4
Participants
  mild adverse events | 1 | 3 | 3
  moderate adverse events | 1 | 1 | 1
  severe adverse events | 0 | 0 | 1

4. Secondary Outcome: Alcohol Craving
Description: Alcohol craving will be measured during Alcohol Drinking Paradigm (ADP) sessions 1, 2 and 3 using the total score of the Alcohol Urge Questionnaire (AUQ). The AUQ has 8 items. Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7; items 2 and 7 are reverse scored). Higher scores reflect greater craving. Total score range is from a minimum of 8 to a maximum of 56. The AUQ is administered before study medication and at various times after study medication. The AUQ score reported here is the highest AUQ score following administration of study medication.
Time Frame: 3 days (1 day each for ADP Session 1, 2, and 3. Each ADP Session included 1 dose of the drug intervention, either Placebo, Lacosamide 100 mg, or Lacosamide 200 mg).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lacosamide 100 mg | Lacosamide 200 mg
Number analyzed (Participants) | 3 | 3 | 4
score on a scale | 34.7 (19.1) | 36 (16.4) | 37.8 (8.9)

5. Secondary Outcome: Alcohol Consumption (Number of Standard Drinks Consumed)
Description: Alcohol consumption is measured during each of the Alcohol Drinking Paradigm (ADP) sessions, 1, 2 and 3. In each session participants received one of the 3 drug interventions, Placebo, Lacosamide 100 mg, or Lacosamide 200 mg. Consumption was measured using the number of alcoholic standard drinks consumed during the ADP sessions. A standard drink per NIAAA definition is 14 grams of pure alcohol.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Placebo | Lacosamide 100 mg | Lacosamide 200 mg
Number analyzed (Participants) | 3 | 3 | 4
standard drinks | 3.44 (2.41) | 2.84 (2.00) | 4.46 (2.83)

6. Secondary Outcome: Subjective Effects of Alcohol Consumption
Description: Subjective effects of alcohol consumption are measured during the Alcohol Drinking Paradigm (ADP) sessions 1, 2 and 3 using the Biphasic Alcohol Effects Scale (BAES), which has 2 subscales; the Stimulation Subscale range is 0 - 70, where 0 is the least and 70 is the greatest stimulation; the Sedation Subscale range is 0 - 70, where 0 is the least and 70 is the greatest sedation. The BAES was administered both before and at various timepoints after study medication administration in each of the ADP sessions. The BAES scores reported here are the peak Stimulation scores after medication administration and peak Sedation scores after medication administration for each of ADP sessions 1, 2 and 3.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Lacosamide 100 mg | Lacosamide 200 mg
Number analyzed (Participants) | 3 | 3 | 4
score on a scale
  Stimulation subscale | 31.3 (27.7) | 44.3 (22.4) | 45.2 (16.0)
  Sedative subscale | 27.3 (4.7) | 26.7 (7.0) | 30.5 (10.0)

ADVERSE EVENTS:
Time Frame: Starting at baseline and ending at follow-up for a total of 5 weeks.
Arm/Group | Placebo | Lacosamide 100 mg | Lacosamide 200 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 3/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Lacosamide 100 mg (N=3) | Lacosamide 200 mg (N=4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Double Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Sensation of spinning (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Sleepiness (General disorders) | 1 (1) | 3 (3) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Loss of coordination of muscle movements (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1 participant withdrew prior to ADP Session 3 and therefore did not receive the drug intervention of Lacosamide 100 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03897348/Prot_SAP_ICF_000.pdf